CLINICAL TRIAL: NCT03282149
Title: A Placebo-controlled, Preliminary Evaluation of Safety, Tolerability, and Efficacy of Ascending Doses of XT-150 for the Treatment of Osteoarthritic Pain
Brief Title: Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xalud Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XT-150-1-0201
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis, Knee
Keywords: inflammation; cytokine; anti-inflammatory; pain
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation; Pain

STUDY DESIGN:
Intervention Model Description: Inflammation and pain due to osteoarthritis in the knee
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unblinded pharmacy provides injection preparation for blinded administration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Dose 1 (Experimental): Lowest trial dose of XT-150
  Interventions: Biological: XT-150
- Dose 2 (Experimental): Second, escalating dose of XT-150
  Interventions: Biological: XT-150
- Dose 3 (Experimental): Third, escalating dose of XT-150
  Interventions: Biological: XT-150
- Saline placebo (Placebo Comparator): 2 of 8 participants in each cohort will randomly be assigned to placebo
  Interventions: Biological: XT-150

INTERVENTIONS:
Biological: XT-150 — IL-10 transgene DNA plasmid injected into the knee synovial capsule

SUMMARY:
Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain - Dose escalation

DETAILED DESCRIPTION:
Preliminary Evaluation of Safety, Tolerability, and Efficacy of XT-150 for the Treatment of Osteoarthritic Pain.

Subjects for whom replacement knee surgery is recommended will be enrolled in the study. A single injection of a DNA plasmid with a variant Interleukin-10 (IL-10) transgene will be injected into the synovial capsule of the knee.

This is a first in human, dose-range, safety and efficacy study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, between 18 and 90 years of age, inclusive. Women who are not of child-bearing potential in the same age range.
2. Sufficiently severe OA of knee to require/have recommended knee replacement surgery or be unsuitable for knee replacement surgery or be unsuitable for knee replacement surgery based on co-morbidities or orthopedic considerations; be free of local or intra-articular infection.
3. Symptomatic disease because of osteoarthritis, defined as one or more of the following Verbal Numerical Rating Scale (VNRS) scores:

   1. a worst pain of at least 7 at any time during the preceding week (based on scale of 0 to 10, with 10 representing "pain as bad as you can imagine").
   2. a worst stiffness of at least 7 at any time during the preceding week (based on a scale of 0 to 10, with 10 representing "stiffness as bad as you can imagine").
4. Stable analgesic regimen during the 4 weeks prior to enrollment.
5. Inadequate pain relief (mean >5 mean on Brief Pain Inventory-Severity Scale) from prior therapies lasting 3 months.
6. In the judgment of the Investigator, acceptable general medical condition
7. Life expectancy >6 months
8. Male participants who are heterosexually active and not surgically sterile must agree to use effective contraception, including abstinence, for the duration of the study and for 3 months after the study is completed.
9. Have suitable knee joint anatomy for intra-articular injection
10. Willing and able to return for the follow-up (FU) visits
11. Able to reliably provide pain assessment
12. Able to read and understand study instructions, and willing and able to comply with all study procedures

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of the study drug, including double-stranded DNA, mannose, and sucrose
2. Scheduled knee replacement within 4 months; participant agrees not to schedule a knee replacement appointment within 4 months of study treatment
3. History of rheumatoid arthritis of the knee
4. High peri-operative risks which in the judgment of the investigator preclude a safe knee injection procedure (e.g., poorly controlled diabetes, cardiac inadequacy such as NYHA class > II, G4 glomerular filtration rate [eGFR < 30 mL/min by Cockcroft-Gault])
5. Current treatment with immunosuppressive (systemic corticosteroid therapy [equivalent to >10mg/day prednisone] or other strong immunosuppressant)
6. History of immunosuppressive therapy; high-potency systemic steroids in the last 3 months.
7. Currently receiving systemic chemotherapy or radiation therapy for malignancy
8. Clinically significant hepatic disease as indicated by clinical laboratory results ≥3 times the upper limit of normal for any liver function test (e.g., aspartate aminotransferase, alanine aminotransferase, lactate dehydrogenase)
9. Severe anemia (Grade 3; hemoglobin <8.0 g/dL, <4.9 mmol/L, <80 g/L; transfusion indicated), uncontrolled coagulopathy (Grade 1, prolonged activated partial prothrombin time (aPTT) > upper limit of normal (ULN) to 1.5xULN), or bleeding diathesis, Grade 1 white cell counts (lymphocytes <LLN - 800/mm3; <LLN - 0.8 x 10e9 /L, neutrophils <LLN - 1500/mm3; <LLN - 1.5 x 10e9 /L)
10. Positive serology for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus within 4 weeks of commencing the study
11. Significant neuropsychiatric conditions; dementia, major depression, or altered mental state that in the opinion of the Investigator will interfere with study participation
12. Current treatment with systemic antibiotics or antivirals (EXCEPTION: topical treatments)
13. Current treatment with anticoagulants, other than low-dose aspirin, prescribed for new onset of symptoms in 3 months before screening visit.
14. Known or suspected history of active alcohol or intravenous/oral drug abuse within 1 year before the screening visit
15. Women of child-bearing potential
16. Use of any investigational drug or device within 1 month before enrollment or current participation in a trial that included intervention with a drug or device; or currently participating in an investigational drug or device study.
17. Any condition that, in the opinion of the Principal Investigator, could compromise the safety of the participant, the participant's ability to communicate the study staff, or the quality of the data

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-21 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety] | 180 days post treatment
  Clinical Pathology, Adverse Events

SECONDARY OUTCOMES:
Verbal Numerical Rating Scale | 180 days post treatment
  0 - 10 Pain assessment

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rickman, MD, Principal Investigator — University of Adelaide
Locations (1):
- CMAX Clinical Research Pty Ltd in collaboration with University of Adelaide, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No
All data will be de-identified in a clinical trial database